CLINICAL TRIAL: NCT00679471
Title: The Relationship Between Early Brain Structure and Development in Full-Term and Pre-Term Infants
Brief Title: Brain Structure and Development in Pre-Term and Full-Term Infants
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Sponsor
Other Study IDs: CCC27122
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: pre-term infants; full-term infants; MRI; brain structure development; pre term; full term
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-Term: Infants born pre-term with birthweight less than 1KG
- Full-Term Infants: Well infants who are born full-term

SUMMARY:
The purpose of this study is to see how full-term and pre-term infants' brains relate to their movement and development throughout the first two years of life. All infants who participate in this study will have a magnetic resonance image (MRI) of the brain prior to discharge from the hospital. Infants will then have follow-up appointments every 3-6 months at home or at the Infant Motor Behavior Laboratory at the University of Delaware. The follow-up sessions will test how infants change their movements to respond to interesting objects or sounds in their environment. It is hoped that the results of this study will assist clinicians in developing better testing and treatment methods for those infants at risk for developmental problems.

ELIGIBILITY:
Inclusion Criteria:

* Pre-term infants (< 1 Kg Birthweight)
* Full-term infants (well)

Max Age: 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pre-term or full-term infants who are admitted to the Neonatal Intensive Care Unit (NICU) at Christiana Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To compare the learning and coordination impairments of extremely low birth weight infants with full term infants at 3 and 6 months of age | 6 months
  To compare the learning and coordination impairments of extremely low birth weight infants with full term infants at 3 and 6 months of age. This is accomplished through a series of play activities.

SECONDARY OUTCOMES:
To relate the learning and coordination impairments of extremely low birth weight infants at 3 and 6 months of age to their CNS impairments at term age. | 6 months
  To relate the learning and coordination impairments of extremely low birth weight infants at 3 and 6 months of age to their CNS impairments at term age.

OTHER OUTCOMES:
To determine the ability of data from learning and coordination impairments and brain MRI / MRS (magnetic resonance spectroscopy) to predict results from common clinical assessments from 3-24 months. | 24 months.
  To determine the ability of data from learning and coordination impairments and brain MRI / MRS (magnetic resonance spectroscopy) to predict results from common clinical assessments from 3-24 months. MRI / MRS (magnetic resonance spectroscopy) of the brain was performed as close to term equivalent age as possible.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Paul, MD, Principal Investigator — Christiana Hospital
Locations (2):
- United States (2):
  - University of Delaware: Infant Motor Beahvior Lab, Newark, Delaware
  - Christiana Hospital, Newark, Delaware

REFERENCES:
- [Derived] Gadin E, Lobo M, Paul DA, Sem K, Steiner KV, Mackley A, Anzilotti K, Galloway C. Volumetric MRI and MRS and early motor development of infants born preterm. Pediatr Phys Ther. 2012 Spring;24(1):38-44. doi: 10.1097/PEP.0b013e31823e069d. PMID 22207464